CLINICAL TRIAL: NCT01900184
Title: Part 1: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Ascending Single Dose and Food Influence Study of QGC001 Administered Orally To Healthy Adult Subjects, Part 2: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Ascending Multiple Dose Study of QGC001 Administered Orally To Healthy Adult Subjects.
Brief Title: Study of the Product QGC001 as a Single Dose and Multiple Doses Administered Orally to Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quantum Genomics SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: QGC001/1QG2
Record Dates: First submitted 2013-06-27; First posted 2013-07-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 500 mg bid of QGC001 (Experimental): Each dose of QGC001 will be administered in solution with 200 mL of purified water.
  Interventions: Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
- 750 mg bid of QGC001 (Experimental): Each dose of QGC001 will be administered in solution with 200 mL of purified water.
  Interventions: Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
- 1,000 mg bid of QGC001 (Experimental): Each dose of QGC001 will be administered in solution with 200 mL of purified water.
  Interventions: Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
- Placebo (Placebo Comparator): The placebo will be administered in solution with 200 mL of purified water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
  Arms: 1,000 mg bid of QGC001; 500 mg bid of QGC001; 750 mg bid of QGC001
Drug: Placebo — Contains magnesium stearate, silica dental type, anhydrous lactose
  Arms: Placebo

SUMMARY:
1QG2 is a Phase 1 study aiming to assess the safety and tolerability of ascending single/multiple oral doses (SAD & MAD) in healthy young subjects, the preliminary food interaction and the effect of QGC001 on blood pressure and heart rate, but also to determine pharmacokinetic preliminary profiles of QGC001 and its metabolite EC33 and pharmacodynamic preliminary profiles of QGC001 and its metabolite EC33 especially effects on the renin-angiotensin-aldosterone and copeptin systems.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian, male healthy subjects of 18 to 45 years of age (inclusive).
* Body weight ≥50 kg, with a body mass index calculated as weight in kg/(height in m2) from 18 to 27 kg/m2 at screening.
* Subjects will sign and date an informed consent form before any study-specific screening procedure is performed.
* Healthy, as determined by the investigator on the basis of medical history, physical examination findings, clinical laboratory test results, vital sign measurements, and digital 12 lead ECG readings.
* Non-smoker or smoker of fewer than 5 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.
* Have a high probability for compliance with and completion of the study.

Exclusion Criteria:

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatological, haematological, neurologic, psychiatric disease or history of any clinically important drug allergy.
* Acute disease state within 7 days before study day 1.
* History of drug abuse within 1 year before study day 1.
* History of alcoholism within 1 year before day 1. Consumption of more than 50 g of ethanol per day.
* Positive serologic findings for human immunodeficiency virus antibodies, hepatitis B surface antigen, and/or hepatitis C virus antibodies.
* Positive findings of urine drug screen (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, MDMA)
* History of any clinically important drug allergy.
* Prohibited Treatments: use of any investigational drug within 90 days or prescription drug within 30 days before investigational medical product administration.
* Consumption of any caffeine-containing products in excess of 6 cups per day (or equivalent), of grapefruit, grapefruit-containing products, or alcoholic beverages within 24 hours before study day 1.
* Use of any over-the-counter drugs including herbal supplements (except for the occasional use of acetaminophen [paracetamol], aspirin and vitamins ≤100% recommended daily allowance) within 7 days before investigational medicinal product administration.
* Donation of blood (i.e. 450 ml) within 90 days before study day 1.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Adverse events | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Red blood cell count | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Haemoglobin | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Haematocrit | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
White blood cell count with differential | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Platelet count | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma sodium | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma potassium | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma calcium | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma total bilirubin | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma conjugated bilirubin | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma Aspartate Amino Transferase (ASAT) | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma Alanine Amino Transferase (ALAT) | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma Gamma Glutamyl Transferase (GGT) | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma alkaline phosphatases | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma total protein | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma Creatine PhosphoKinase (CPK) | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma creatinine | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma glucose | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma cholesterol | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Plasma triglycerides | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Urinary pH | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Urinary protein | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Urinary glucose | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Urinary leukocytes | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Urinary nitrites | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Urinary ketones | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Urinary blood | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Weight assessment (kg) | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Body temperature (°C) | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Supine and orthostatic (systolic and diastolic) blood pressure | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
Heart rate | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD
12-lead ECG | up to 4 weeks for SAD, 5 weeks for FI and 6 weeks for MAD

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of QGC001 | up to 3 days for SAD and FI, up to 9 days for MAD
  Cohorts SAD 1 to 4 and MAD 1 to 3.
Time at which Cmax is observed (tmax) of QGC001 | up to 3 days for SAD and FI, up to 9 days for MAD
  Cohorts SAD 1 to 4 and MAD 1 to 3.
Elimination rate constant (λz) of QGC001 | up to 3 days for SAD and FI, up to 9 days for MAD
  Cohorts SAD 1 to 4 and MAD 1 to 3.
Terminal half-life (t1/2,z) of QGC001 | up to 3 days for SAD and FI, up to 9 days for MAD
  Cohorts SAD 1 to 4 and MAD 1 to 3.
Area Under the Concentration-time curve (AUClast and AUC0-∞) of QGC001 | up to 3 days for SAD and FI, up to 9 days for MAD
  Cohorts SAD 1 to 4 and MAD 1 to 3.
Maximum observed plasma concentration (MRCmax) of metabolic ratios | up to 3 days for SAD and FI, up to 9 days for MAD
  Cohorts SAD 1 to 4 and MAD 1 to 3.
Area Under the Concentration-time curve (MRAUC) of metabolic ratios | up to 3 days for SAD and FI, up to 9 days for MAD
  Cohorts SAD 1 to 4 and MAD 1 to 3.
Cumulative amount eliminated (Ae) | up to 2 days for SAD and FI, up to 8 days for MAD
  Cohorts SAD 1 to 4 and MAD 1 to 3.
Fraction recovered (Fe) | up to 2 days for SAD and FI, up to 8 days for MAD
  Cohorts SAD 1 to 4 and MAD 1 to 3.
Renal clearance (CLR) | up to 2 days for SAD and FI, up to 8 days for MAD
  Cohorts SAD 1 to 4 and MAD 1 to 3.
Plasma renin | up to 2 days for SAD and FI, up to 8 days for MAD
  Determination of renin in blood samples. Cohorts SAD 1 to 3 and MAD 1 to 3.
Plasma aldosterone | up to 2 days for SAD and FI, up to 8 days for MAD
  Determination of aldosterone in blood samples. Cohorts SAD 1 to 3 and MAD 1 to 3.
Plasma cortisol | up to 2 days for SAD and FI, up to 8 days for MAD
  Determination of cortisol in blood samples. Cohorts SAD 1 to 3 and MAD 1 to 3.
Plasma copeptin | up to 2 days for SAD and FI, up to 8 days for MAD
  Determination of copeptin in blood samples. Cohorts SAD 1 to 3 and MAD 1 to 3.
Urinary aldosterone | up to 2 days for SAD and FI, up to 8 days for MAD
  Aldosterone analysis in urine samples. Cohorts SAD 1 to 3 and MAD 1 to 3.
Urinary cortisol | up to 2 days for SAD and FI, up to 8 days for MAD
  Cortisol analysis in urine samples. Cohorts SAD 1 to 3 and MAD 1 to 3.
Urinary sodium | up to 2 days for SAD and FI, up to 8 days for MAD
  Sodium analysis in urine samples. Cohorts SAD 1 to 3 and MAD 1 to 3.
Urinary potassium | up to 2 days for SAD and FI, up to 8 days for MAD
  Potassium analysis in urine samples. Cohorts SAD 1 to 3 and MAD 1 to 3.
Urinary creatinine | up to 2 days for SAD and FI, up to 8 days for MAD
  Creatinine analysis in urine samples. Cohorts SAD 1 to 3 and MAD 1 to 3.
Systolic and Diastolic Blood Pressure | up to 8 days for MAD
  Cohorts MAD 1 to 3.
Heart Rate | up to 8 days for MAD
  Cohorts MAD 1 to 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial PARIS, Rueil-Malmaison, France

REFERENCES:
- [Derived] Khosla J, Aronow WS, Frishman WH. Firibastat: An Oral First-in-Class Brain Aminopeptidase A Inhibitor for Systemic Hypertension. Cardiol Rev. 2022 Jan-Feb 01;30(1):50-55. doi: 10.1097/CRD.0000000000000360. PMID 33027067